CLINICAL TRIAL: NCT04472975
Title: Disease-modifying Drug Safety and Effectiveness in Multiple Sclerosis [DRUMS]
Brief Title: Prescription Drug Safety and Effectiveness in Multiple Sclerosis
Acronym: DRUMS
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: University of Manitoba (Other); Dalhousie University (Other); University of Saskatchewan (Other); Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Helen Tremlett, Professor, Canada Research Chair in Neuroepidemiology and Multiple Sclerosis, University of British Columbia
Other Study IDs: H18--00407; CIHR PJT-156363 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); CIHR FDN-159934 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2020-07-03; First posted 2020-07-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: disease-modifying drugs; health administrative data; population-based; Canada; cohort studies
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis (MS) cohort: Individuals with multiple sclerosis without any exposure to disease-mofidying drugs (DMDs) and with exposure to one or more DMDs.
  Interventions: Drug: Exposure to one or more disease-modifying drug(s)(DMDs) used to treat MS

INTERVENTIONS:
Drug: Exposure to one or more disease-modifying drug(s)(DMDs) used to treat MS — Individuals with MS exposed to one or more DMDs (beta-interferon, glatiramer acetate, natalizumab, fingolimod, dimethyl fumarate, teriflunomide, alemtuzumab, daclizumab or ocrelizumab; regardless of dose, frequency or duration of treatment) between 1st January 1996 and 31st March 2018 in five Canadian provinces.

SUMMARY:
The goal of our research is to find out how safe and effective the drugs used to treat multiple sclerosis (MS) are when used in the everyday, real world. To achieve these study goals, we have two main study Themes. The first Theme focuses on how effective the MS drugs are. We will examine whether the MS drugs can extend life expectancy or prolong a person's ability to stay mobile and walk. We will also look at whether the MS drugs have a beneficial effect on reducing the number of times a person with MS is admitted to a hospital or visits a physician. The second Theme focuses on side effects, including whether the MS drugs are associated with harmful effects, such as cancer, stroke or depression. We will be able to compare the different MS drugs to each other. Also, we will see if men and women or people of different ages and with other illnesses (such as having both MS and diabetes) respond to the MS drugs differently. Our findings will help people with MS and their physicians when trying to make decisions as to which MS drug might be best for them.

DETAILED DESCRIPTION:
Study population:

A validated case definition of multiple sclerosis (MS) will be applied to the health administrative data to identify all MS patients in 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan and Alberta; Studies 1,2,4-6). Developed in Manitoba, the positive predictive value was 80.5% and negative predictive value (NPV) was 75.5% among a population of persons with ≥1 claim for any demyelinating disease. The NPV would be >99% at the general population level where more than 98% of individuals have no claims for demyelinating disease. The algorithm has been successfully applied in British Columbia, Nova Scotia and Saskatchewan.

When MS-specific clinical data are used (British Columbia, Manitoba, Nova Scotia; Study 3), the diagnosis is neurologist confirmed, according to the prevailing international criteria.

Study period:

The earliest study start is Jan/1996 (the 1st full year that DMDs were available and the first year of available administrative and DMD-related data), and the latest study end is March 31, 2018; this represents >2 decades of drug and patient-related follow-up.

Study entry:

Most recent of 1-Jan-1996, an individual's 18th birthday, date of 1st MS-related claim or date of 1st MS clinic visit (when clinical data are accessed [Study 3]).

Study end:

Earliest of death, emigration from the respective province, last MS clinic visit (when clinical data are accessed [Study 3]), or 31-December-2017 (British Columbia, Manitoba, Nova Scotia, Alberta) or 31-March-2018 (Saskatchewan).

DMD exposure:

DMD use, as identified using prescription data. An individual's exposure status can change over time and will be dynamically classified as: 1) no DMD, 2) any DMD, then by generation: 2a) any 1st or 2b) 2nd generation DMD. When possible, the individual drug classes will be explored (beta-interferon [as one class], glatiramer acetate, natalizumab, fingolimod, dimethyl fumarate, teriflunomide, alemtuzumab).

Time perspective:

Analyses of prospectively recorded health administrative, prescription and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* All MS patients (Studies 1, 2, 4-6) who have resided in one of the 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan or Alberta) over the study period as identified using a validated case definition of MS that will be applied to health administrative data (≥ 3 records related to MS coded during physician or hospital visits, or prescription filled for a MS-specific DMDs).
* Subjects require 1 year of residency in a province before study entry to enable sufficient data to facilitate covariate creation, e.g. comorbidity, and to identify those with prior DMD use.
* All adults who visited a MS clinic in British Columbia, Manitoba or Nova Scotia (Study 3), were diagnosed with MS and had a relapsing-onset disease course and at least one EDSS score of 6.5 or less, recorded on or after: January 1st 1996 (British Columbia) or April 1st 1996 (Manitoba) or January 1st 1998 (Nova Scotia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A MS cohort study (Studies 1, 2, 4-6) will be identified using a validated case definition of MS that will be applied to the whole-population linked administrative health data in five Canadian provinces spanning from west to east coast: British Columbia (BC; population 4.65 million [2016]), Alberta (AB; 4.07 million population [2016]), Saskatchewan (SK; population 1.10 million [2016]), Manitoba (MB; population 1.28 million [2016]) and Nova Scotia (NS; population 924,000 [2016]).
  When MS-specific clinical data are used (British Columbia, Manitoba, Nova Scotia; Study 3), the diagnosis is neurologist confirmed, according to the prevailing international criteria.
  Within each province, we anticipate finding virtually the whole population of people living with MS via the administrative data, and, in the clinical data, ≈60-80% or 100% of those seeking DMDs (the MS clinics are the sole prescribers of the DMDs).
Sampling Method: Probability Sample
Enrollment: 35000 (Actual)
Dates: Start 1996-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Study 1: All-cause hospitalizations | As recurrent events from study entry to study end, up to 22 years.
  The outcome (all-cause hospitalizations) will be derived from the comprehensive hospital data, excluding pregnancy-related events, in 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan and Alberta).
Study 2: All-cause mortality | Measured using Cox proportional hazards models (time from study entry to death), up to 22 years.
  The outcome (all-cause mortality) will be derived from the province-wide death data (e.g., Vital Statistics or the equivalent) in 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan and Alberta).
Study 3: Change in disability (Expanded Disability Status Scale [EDSS]) over time | Assessed using mixed effects model from study entry to study end, up to 22 years.
  The outcomes (change in EDSS) will be derived from the MS clinical data in 3 Canadian provinces (British Columbia, Manitoba and Nova Scotia).

SECONDARY OUTCOMES:
Study 1: Physician consultation rates (overall and by physician specialty) | Overall numbers of physician consultations will be measured from study entry to study end, up to 22 years of follow-up.
  The outcome (physician consultation) will be derived from the physician data, excluding pregnancy-related events, in 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan and Alberta).
Study 3: MS disability, measured using the Expanded Disability Status Scale (EDSS) and assessed as time to sustained EDSS 6 | Measured using Cox proportional hazards models (time from study entry to sustained EDSS 6 confirmed after at least 6 months with no subsequent improvement), up to 22 years of follow-up.
  The outcome (sustained EDSS 6) will be derived from the MS clinical data in 3 Canadian provinces (British Columbia, Manitoba and Nova Scotia).
Study 3: Sustained EDSS 4 | Measured using Cox proportional hazards models (time from study entry to sustained EDSS 4), up to 22 years of follow-up.
  The outcomes (sustained EDSS 4) will be derived from the MS clinical data in 3 Canadian provinces (British Columbia, Manitoba and Nova Scotia).
Study 4: Explore the modifying effects | From study entry to study end, up to 22 years of follow-up.
  Effects of sex, age, comorbidity and DMD treatment duration on outcomes (all-cause hospitalizations, physician consultation rates, all-cause mortality, changes in EDSS) will be assessed.
Study 5: Potential incident adverse events | Time from study entry to the incident adverse event of interest will be assessed using Cox proportional hazards with time-varying DMD exposure, up to 22 years of follow-up.
  'Incident' event defined as not present in the year before DMD initiation. The outcomes (incident adverse events) will be identified using physician and hospital claims, coded using International Classification of Diseases [ICD]-9/10 and prescriptions filled (by ATC levels), in 5 Canadian provinces (British Columbia, Manitoba, Nova Scotia, Saskatchewan and Alberta). An additional, data mining, discovery approach will assess the associations between exposure and adverse events using unsupervised machine learning techniques. Cases of PML will be described.
Study 6: Characteristics associated with risk of adverse events | From study entry to study end, up to 22 years of follow-up.
  Examine demographic and clinical characteristics associated with risk of adverse events, including sex, age, comorbidity and DMD treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Tremlett, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No
The data that were used for this study reside on a limited access secure research environment and for legal and ethical reasons, the data cannot leave this secure research environment. However, researchers can apply to access the health administrative data held within each province.

REFERENCES:
- [Derived] Ng HS, Zhu F, Kingwell E, Zhao Y, Yao S, Ekuma O, Svenson LW, Evans C, Fisk JD, Marrie RA, Tremlett H. Disease-modifying drugs for multiple sclerosis and subsequent health service use. Mult Scler. 2022 Apr;28(4):583-596. doi: 10.1177/13524585211063403. Epub 2021 Dec 24. PMID 34949130